CLINICAL TRIAL: NCT00486681
Title: Evaluation of the Implementation of the Accu-Chek Inform Cobas IT 1000 System in Three Medical Hospital Departments: Impact on the Management of Diabetes
Brief Title: Clinical Assessment of an in-Patient Glucose Monitoring System (Accu-Chek Inform Cobas IT 1000)
Acronym: COBAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Roche Diagnostics Meylan France (Unknown); Assistance Medico-Technique A Domicile (Other)
Responsible Party: Nelly Wion, University Hospital of Grenoble
Other Study IDs: DCIC 05 51
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2008-02

CONDITIONS: Diabetes Mellitus; Blood Glucose; Hospital Information Systems; Medical Device
Keywords: Glucose monitoring; Diabetes management; Information system; In-patient glycemic control
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: period I (warning of the Accu-Check Inform glucose meter on glucose levels not activated)
- 2: period II (warning activated).
  Interventions: Device: Accu Chek Inform and Cobas IT 1000

INTERVENTIONS:
Device: Accu Chek Inform and Cobas IT 1000 — period II (warning activated)
  Other Names: Accu Chek Inform
  Groups: 2

SUMMARY:
The principal objective of this single-center 2-period study is to evaluate the glycemic control of in-patients in 3 hospital departments (Diabetology, Cardiology and Pulmonary Care) as the rate of capillary blood glucose measurements within a pre-define target range, and to compare results during the period I (warning of the Accu-Check Inform glucose meter on glucose levels not activated) and period II (warning activated).

DETAILED DESCRIPTION:
The study is a 6-month large scale assessment of an information system consisting in a glucose meter with multiple alerts (Accu-Chek Inform) associated with a data base (Cobas IT 1000) in order to share the results of glucose monitoring using the hospital information network.

The appraisal of the glycemic control was based on the rate of capillary blood glucose measurements within a pre-defined target range (3.9-8.5 mMol/l) during each study period.

Whether the system implementation can improve the outcome related to the management of in-patients with diabetes is assessed in 3 hospital departments (Diabetology, Cardiology and Pulmonary Care) as follows:

* principal objective, glycemic control of in-patients (Cardiology and Pulmonary Care) as the rate of capillary blood glucose (CBG) values within the pre-defined target range, and comparison of results observed during period I (meter warning not activated) and period II (warning of the meter on out-of-target glucose level activated).
* the impact on the performance of quality controls of CBG measurements with (period II) or without (period I) activation of a warning on the meter related to inappropriate quality control frequency (all departments).
* evaluate the traceability of CBG results and compare it with (period II) or without (period I) the activation of the automatic record of data ensured by the Accu-Chek Inform meter and Cobas IT 1000 data base (all departments).
* during a sub-period of period II, the impact on patient glycemic control of the intervention of a diabetologist, determined by the activation of a warning sent to the physician in case of out of target CBG results via the Cobas IT 1000 data base (Cardiology and Pulmonary Care).
* the impact of the above warning activation plus diabetologist intervention on the incidence of low CBG.

ELIGIBILITY:
Inclusion Criteria:

* In-patients,
* Age > 18 years,
* Requiring a monitoring of capillary blood glucose levels

Exclusion Criteria:

* No glucose monitoring needed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring a monitoring of capillary blood glucose levels
Sampling Method: Non-Probability Sample
Enrollment: 949 (Actual)
Dates: Start 2007-01; Primary Completion 2007-07 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
compare glycemic control of patients hospitalized in 3 departments | hospitalisation period

SECONDARY OUTCOMES:
number of glycemia controls | hospitalisation period
number of traceable glycemia readings | hospitalisation period
number of hypoglycemia events and frequency of measures taken | hospitalisation period
mean of % of glycemia for patients in warning phase with or without diabetologist intervention | hospitalisation period

CONTACTS AND LOCATIONS:
Overall Officials: NELLY WION, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital of Grenoble, Grenoble, France

REFERENCES:
- [Background] Kucher N, Koo S, Quiroz R, Cooper JM, Paterno MD, Soukonnikov B, Goldhaber SZ. Electronic alerts to prevent venous thromboembolism among hospitalized patients. N Engl J Med. 2005 Mar 10;352(10):969-77. doi: 10.1056/NEJMoa041533. PMID 15758007
- [Background] ACE/ADA Task Force on Inpatient Diabetes. American College of Endocrinology and American Diabetes Association Consensus statement on inpatient diabetes and glycemic control. Diabetes Care. 2006 Aug;29(8):1955-62. doi: 10.2337/dc06-9913. No abstract available. PMID 16873812
- [Background] Inzucchi SE, Rosenstock J. Counterpoint: Inpatient glucose management: a premature call to arms? Diabetes Care. 2005 Apr;28(4):976-9. doi: 10.2337/diacare.28.4.976. No abstract available. PMID 15793210
- [Background] Clement S, Braithwaite SS, Magee MF, Ahmann A, Smith EP, Schafer RG, Hirsch IB; American Diabetes Association Diabetes in Hospitals Writing Committee. Management of diabetes and hyperglycemia in hospitals. Diabetes Care. 2004 Feb;27(2):553-91. doi: 10.2337/diacare.27.2.553. No abstract available. PMID 14747243
- [Background] Halimi S. [Benefits of blood glucose self-monitoring in the management of insulin-dependent (IDDM) and non-insulin-dependent diabetes (NIDDM). Analysis of the literature: mixed results]. Diabetes Metab. 1998 Nov;24 Suppl 3:35-41. French. PMID 9881230
- [Background] King H, Aubert RE, Herman WH. Global burden of diabetes, 1995-2025: prevalence, numerical estimates, and projections. Diabetes Care. 1998 Sep;21(9):1414-31. doi: 10.2337/diacare.21.9.1414. PMID 9727886
- [Background] Mise en place et conduite en France d'essais cliniques portant sur des dispositifs médicaux et dispositifs médicaux de diagnostic in vitro.Afssaps September 2006, 15. http://agmed.sante.gouv.fr